CLINICAL TRIAL: NCT00178321
Title: Improving Sleep and Outcomes in Critically Ill Children
Brief Title: Improving Sleep in the Pediatric Intensive Care Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10055
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Critically Ill
Keywords: Sleep; Criticall Ill; Children; Earplugs
MeSH Terms: conditions — Critical Illness | interventions — Ear Protective Devices

INTERVENTIONS:
Device: earplugs

SUMMARY:
Sleep is disrupted in the PICU. This disruption has been reported in studies that have used: (a) observation of sleep-wake cycles (b) self-reports by children themselves , and (c) objective measures (e.g., electroencephalograph( EEG). Noise and light levels have been correlated with profound sleep disruption in the PICU . Sleep disruption is known to have a profound impact on the overall health of a child, both from a physiological and a psychological standpoint . In addition, sleep disruption has been shown to change cortisol levels, cause impaired immune responses and impair cognitive function in both children and adults . Disruption in sleep also is known to impair healing through these many complex connections with other homeostatic processes in the human body. What is the effect of wearing earplugs in critically ill children admitted to the PICU on:

1. Sleep states
2. Physiological stability (e.g. melatonin, cortisol and immune status)
3. Sleep habits after discharge from the PICU (on the general pediatric unit, 2 weeks and 2 months after discharge), and
4. Child behavior at 2 weeks and 2 months after discharge from the PICU by parent report on the Child Behavior Checklist (CBCL).

DETAILED DESCRIPTION:
While often life saving, the need for admission to the pediatric intensive care unit (PICU) places children in a profoundly artificial environment that has the potential to alter the biological processes that defend homeostasis. All living organisms have biological rhythms that serve as their basic organizing feature. These rhythms vary widely, ranging from seconds (e.g., heartbeat) to weeks (menstrual cycle). Biological rhythms that have a 24-hour cycle are termed circadian rhythms. Of the many circadian rhythms, the sleep-wake cycle is the most evident [2]. Other biological processes that have a circadian rhythm include growth hormone, melatonin, and cortisol secretion .

Sleep is disrupted in the PICU. This disruption has been reported in studies that have used: (a) observation of sleep-wake cycles [6, 7]; (b) self-reports by children themselves, and (c) objective measures (e.g., electroencephalograph( EEG). Noise and light levels have been correlated with profound sleep disruption in the PICU . Sleep disruption is known to have a profound impact on the overall health of a child, both from a physiological and a psychological standpoint . In addition, sleep disruption has been shown to change cortisol levels, cause impaired immune responses and impair cognitive function in both children and adults . Disruption in sleep also is known to impair healing through these many complex connections with other homeostatic processes in the human body.

There is a dearth of research on improving sleep and reversing the negative effects of sleep disruption on homeostasis in critically ill children

RQ1: What is the effect of wearing earplugs in critically ill children admitted to the PICU on:

1. Sleep states
2. Physiological stability (e.g. melatonin, cortisol and immune status)
3. Sleep habits after discharge from the PICU (on the general pediatric unit, 2 weeks and 2 months after discharge), and
4. Child behavior at 2 weeks and 2 months after discharge from the PICU by parent report on the Child Behavior Checklist (CBCL).

ELIGIBILITY:
Inclusion Criteria:

* Parents or primary caregivers ages 18 years or older, who can read and speak English and their critically ill children who meet the following criteria will be eligible for participation (a) ages 1-15 years, (b) anticipated survival, (c) no severe handicapping (neurological) conditions, (d) not a prior transplant patient, (e) no active oncology or metabolic process (other than diabetes), (f) not diagnosed with a traumatic brain injury and (a) between 1 and 15 years of age, (b) expected length of stay >2days, (c) expected to live, and (d) parents that can read and write English

Exclusion Criteria:

* diagnosis of cancer, a previous transplant patient, diagnosis of a metabolic disorder (except for diabetes), neurological conditions that would affect sleep wake cycles, a traumatic brain injury patient, evidence of abuse. These conditions are known to affect sleep patterns and/or immune system and (a) not meeting inclusion criteria, (b) anticipated death of the child, (c) parents/primary caregiver make a personal choice to withdraw themselves and their child from the study, (d) the child has evidence of abuse.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-09; Study Completion 2006-08

PRIMARY OUTCOMES:
To pilot test the changes in sleep patterns with the use of earplugs in the PICU

SECONDARY OUTCOMES:
To see if there are neurobehavioral differences in children who use the earplugs in the PICU vs, those who do not

CONTACTS AND LOCATIONS:
Overall Officials: Margaret-Ann Carno, PhD, RN, Principal Investigator — University of Rochester; Heidi V. Connolly, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States